CLINICAL TRIAL: NCT03985865
Title: The Influence of Bitter Substrates on Hunger, Gastrointestinal Hormone Release and Hedonic Food Intake
Brief Title: IG vs ID Bitter Administration
Acronym: IG vs ID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S551166
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-01

CONDITIONS: Obesity
Keywords: Bitter; Motilin; Ghrelin; CCK; GLP-1; SST; Denatonium benzoate; Quinine hydrochloride
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Intragastric quinine hydrochloride (Experimental): 10 µmol of quinine hydrochloride per kg body weight was administrated into the stomach.
  Interventions: Drug: Intragastric quinine hydrochloride
- intragastric denatonium benzoate (Experimental): 1 µmol of denatonium benzoate per kg body weight was administrated into the stomach.
  Interventions: Drug: Intragastric denatonium benzoate
- Intragastric placebo (Placebo Comparator): 0.1 ml of water (placebo) per kg body weight was administrated into the stomach.
  Interventions: Drug: Intragastric placebo
- Intraduodenal quinine hydrochloride (Experimental): 10 µmol of quinine hydrochloride per kg body weight was administrated into the duodenum.
  Interventions: Drug: Intraduodenal quinine hydrochloride
- Intraduodenal denatonium benzoate (Experimental): 1 µmol of denatonium benzoate per kg body weight was administrated into the duodenum.
  Interventions: Drug: Intraduodenal denatonium benzoate
- Intraduodenal placebo (Placebo Comparator): 0.1 ml of water (placebo) per kg body weight was administrated into the duodenum.
  Interventions: Drug: Intraduodenal placebo

INTERVENTIONS:
Drug: Intragastric quinine hydrochloride — A nasogastric feeding tube was positioned into the stomach, and checked with a pH strip. 10 µmol of quinine hydrochloride per kg body weight was administrated into the stomach.
  Other Names: IG QHCl
  Arms: Intragastric quinine hydrochloride
Drug: Intragastric denatonium benzoate — A nasogastric feeding tube was positioned into the stomach, and checked with a pH strip. 1 µmol of denatonium benzoate per kg body weight was administrated into the stomach.
  Other Names: IG DB
  Arms: intragastric denatonium benzoate
Drug: Intragastric placebo — A nasogastric feeding tube was positioned into the stomach, and checked with a pH strip. 0.1 ml of water (placebo) per kg body weight was administrated into the stomach.
  Other Names: IG PLC
  Arms: Intragastric placebo
Drug: Intraduodenal quinine hydrochloride — A nasogastric feeding tube was positioned into the duodenum, and checked with fluoroscopy. 10 µmol of quinine hydrochloride per kg body weight was administrated into the duodenum.
  Other Names: ID QHCl
  Arms: Intraduodenal quinine hydrochloride
Drug: Intraduodenal denatonium benzoate — A nasogastric feeding tube was positioned into the duodenum, and checked with fluoroscopy. 1 µmol of denatonium benzoate per kg body weight was administrated into the duodenum.
  Other Names: IG DB
  Arms: Intraduodenal denatonium benzoate
Drug: Intraduodenal placebo — A nasogastric feeding tube was positioned into the duodenum, and checked with fluoroscopy. 0.1 ml of water (placebo) per kg body weight was administrated into the duodenum.
  Other Names: ID PLC
  Arms: Intraduodenal placebo

SUMMARY:
We want to investigate whether bitter compounds, denatonium benzoate and quinine hydrochloride, have a distinct effect on gastrointestinal hormone release after infusion into the stomach or duodenum. Furthermore, we want to observe an effect on hunger sensations and hedonic food intake. Moreover, we suggest somatostatin as a driving factor for decreased motilin and ghrelin release after intragastric administration.

DETAILED DESCRIPTION:
Intragastric administration of the bitter tastants denatonium benzoate (DB) or quinine hydrochloride (QHCl) decreases orexigenic hormone levels, and reduces hunger sensations. Contradictory, in vitro studies on human gastric and duodenal tissue showed that DB exposure increased motilin and octanoylated ghrelin levels. DB stimulated somatostatin (SST) release, which is an inhibiting paracrine hormone. We hypothesized that the reduction in hunger ratings and hormone levels is stronger after intragastric compared to intraduodenal administration, and that these differences are mediated by differential SST release. Fourteen healthy female volunteers participated in a randomized, placebo-controlled crossover study. After an overnight fast, DB (1 µmol/kg), QHCl (10 µmol/kg) or placebo were given intragastric or intraduodenal via a feeding tube. Blood samples were taken at regular time points to obtain the hormonal release. Hunger was rated at the same points on a 100 mm visual analog scale (VAS). Ad libitum milkshake intake was assessed at the end of the experiment and taste was scored on a VAS.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female between 18 and 65 years of age.
* Subject has a BMI between 18 and 25 kg/m² and has a stable body weight for at least 3 consecutive months at the start of the study and keeps a stable weight during the study visits.
* Women of child-bearing potential agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject is under age of legal consent, male, pregnant or breastfeeding.
* Subject with a BMI ≥ 18 kg/m² or BMI ≤ 25 kg/m².
* Subject has current symptoms or a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies.
* Subject has diabetes.
* Subject has a significant heart, lung, liver or kidney disease.
* Subject has any history of a neurological disorder.
* Subject has a history of abdominal surgery. Those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate.
* Subject shows abnormal eating behavior or has an eating disorder.
* History or current use of drugs that can affect glycaemia, gastrointestinal function, motility or sensitivity or gastric acidity.
* History or current use of centrally acting medication, including antidepressants, antipsychotics and/or benzodiazepines (in the last year before screening visit).
* Subject consumes excessive amounts of alcohol, defined as >14 units per week.
* Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
* High caffeine intake (> 500 ml coffee daily or equivalent).
* Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.
* Recent participation (<30 days) or simultaneous participation in another clinical study.
* Subjects with lactose intolerance.
* Subjects with quinine allergy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female volunteers have a higher chance to be more sensitive for bitter compounds because of their genetic background in comparison to males.
Enrollment: 14 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Changes in plasma levels of motilin, ghrelin, somatostatin, GLP-1 and CCK after bitter administration into the stomach or duodenum | A first blood sample is taken as a reference 10 min before administration of the condition. After the infusion, every 10 min blood samples are taken for 2 hours.
  Infusion of bitter compounds into the stomach or duodenum is performed via a nasogastric feeding tube. Afterwards, an intravenous dwelling line is placed to take blood samples at several time points during the experiment. Hormone levels of motilin, ghrelin, somatostatin, GLP-1 and CCK are collected with according enzyme inhibitors.

SECONDARY OUTCOMES:
Changes in hunger scores after bitter administration into the stomach or duodenum | Hunger is scored every 10 min during the whole experiment starting 20 min before the infusion, until 2 hours after the infusion. 1 minute before and after ad libitum drinking, hunger is scored.
  Infusion of bitter compounds into the stomach or duodenum is performed via a nasogastric feeding tube. Hunger is scored on a 100 mm visual analog scale at several time points during the experiment. Two hours after the infusion, the nasogastric feeding tube and intravenous dwelling line are removed and the subject drinks ad libitum from a chocolate milkshake until they are fully satisfied. Hunger is scored right before and after drinking the milkshake.
Changes in hedonic food intake after bitter administration into the stomach or duodenum | 2 hours after the infusion of a condition, subjects drink from the milkshake without an intermission.
  Infusion of bitter compounds into the stomach or duodenum is performed via a nasogastric feeding tube. Two hours after the infusion of a bitter compound or placebo, the subjects drink ad libitum from a chocolate milkshake until they are fully satisfied. The milkshake is weighted before and after the experiment to calculate the amount of consumed calories (1 g milkshake = 1 kcal).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — UZ Leuven
Locations (1):
- TARGID, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Verbeure W, Deloose E, Toth J, Rehfeld JF, Van Oudenhove L, Depoortere I, Tack J. The endocrine effects of bitter tastant administration in the gastrointestinal system: intragastric versus intraduodenal administration. Am J Physiol Endocrinol Metab. 2021 Jul 1;321(1):E1-E10. doi: 10.1152/ajpendo.00636.2020. Epub 2021 May 24. PMID 34029163